CLINICAL TRIAL: NCT01207453
Title: Milnacipran in the Treatment of Widespread, Non-Joint Pain in Rheumatoid Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Forest Laboratories (Industry); National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Yvonne C. Lee, Yvonne C. Lee, MD, MMSc, Brigham and Women's Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAV-MD-16; K23AR057578 (NIH)
Record Dates: First submitted 2010-09-21; First posted 2010-09-23 (Estimated); Results first posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Arthritis, Rheumatoid
Keywords: Arthritis, Rheumatoid; Milnacipran; Pain
MeSH Terms: conditions — Arthritis, Rheumatoid; Pain | interventions — Milnacipran

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Milnacipran then placebo (Other): This arm of the study will contain half the study population after randomization. The participants in this arm will receive milnacipran for 6 weeks. They will undergo a one-week taper and a two week washout period and then crossover to a placebo for 6 weeks.
  Interventions: Drug: Milnacipran; Drug: Placebo
- Placebo then milnacipran (Other): This arm of the study will contain half the study population after randomization. The participants in this arm will receive placebo for 6 weeks. They will undergo a one-week "taper" and a two week "washout" period and then crossover to milnacipran for 6 weeks.
  Interventions: Drug: Milnacipran; Drug: Placebo

INTERVENTIONS:
Drug: Milnacipran — Milnacipran comes in 50 mg tablets and is taken orally. Participants will gradually be increased to a target dose of 50 mg twice daily.
  Other Names: Savella
Drug: Placebo

SUMMARY:
The purpose of this study is to determine whether milnacipran reduces widespread, non-joint pain in patients with rheumatoid arthritis (RA). The investigators will conduct a double-blind randomized crossover trial in subjects with RA to test the hypothesis that milnacipran improves widespread, non-joint pain. The investigators will also use data from the trial to determine whether response to milnacipran is associated with pain-modulating mechanisms from the central nervous system. The investigators hypothesize that response to milnacipran will be greater among patients with impaired central pain mechanisms than among patients with intact central pain modulating mechanisms.

DETAILED DESCRIPTION:
Despite the development of effective medications to treat inflammation, pain remains a priority for rheumatoid arthritis (RA) patients. The pain that persists despite anti-inflammatory treatment is usually widespread and non-articular; it may lead to diminished quality of life and high medical, psychological and social costs. To develop better treatments for pain and prevent disability, it is critical to obtain a better understanding of widespread, non-joint pain in RA.

Milnacipran is a selective serotonin-norepinephrine reuptake inhibitor (SNRI). No studies have examined the effect of SNRIs on pain in RA. However, several studies have examined the role of SNRIs in fibromyalgia and related pain conditions. Treatment with milnacipran has been associated with improvements in clinical pain severity in Phase 2 and Phase 3 randomized placebo-controlled trials of fibromyalgia patients. In animal models, milnacipran appears to moderate the pain-inducing effects of inflammation and central sensitization. Thus milnacipran may be an ideal drug to treat pain in RA.

A clinical trial of an SNRI in the treatment of widespread, non-joint pain in RA will provide more information regarding pain mechanisms and may lead to more targeted, effective ways of treating pain in RA.

ELIGIBILITY:
Inclusion Criteria:

* Age 24 years or older
* Primary diagnosis of rheumatoid arthritis from a board-certified rheumatologist
* Willing to maintain stable doses of concurrent non-steroidal anti-inflammatory drugs or other acceptable medications or therapies for the duration of the study
* Brief Pain Inventory Average Pain >= 4 at the screening visit
* Widespread Pain Index >= 5 at the screening visit
* Able to give informed consent

Exclusion Criteria:

* Diagnosis of primary fibromyalgia
* Diagnosis of cold sensitive conditions such as Raynaud's syndrome, cryoglobulinemia and paroxysmal cold hemoglobinuria
* Diagnosis of psychotic disorders, such as schizophrenia, schizoaffective disorder, delusional disorder and shared psychotic disorder
* Patients being treated with SSRIs, MAO inhibitors or tricyclic, tetracyclic or atypical antidepressants for pain may participate in this study if they are washed off these medications before study entry. Patients currently receiving therapy with SSRIs or tricyclic, tetracyclic or atypical antidepressants for depression may be washed off these medications before study entry pending permission of the prescribing physician and if they have never received a diagnosis of major depressive disorder or had a history of suicidal ideation.
* Patients on thioridazine or MAO inhibitors
* Patients taking codeine or other opioids/opiates. Patients who are taking medications such as pregabalin (Lyrica) and gabapentin (Neurontin) for pain may be enrolled in this study.
* Known hypersensitivity to milnacipran
* Patients with a significant risk of suicide as assessed by the Beck depression inventory form
* Patients with a history of suicide
* Pregnant or breast-feeding women
* Patients with an actively pending worker's compensation claim or auto no-fault claim; patients with current worker's compensation, auto no-fault compensation, or litigation; or any patient with significant secondary gain issues per discretion of the researchers.
* Patients with myocardial infarction within the past 12 months, active cardiac disease (chest pain or evidence of ischemia on stress test), acute congestive heart failure requiring hospitalization in the past 12 months, clinically significant cardiac rhythm or conduction abnormalities requiring hospitalization in the past 12 months
* Patients with severe liver impairment (AST or ALT > 3 times the upper limit of normal)

  * For patients 2-3 times the upper limit of normal, we will obtain enrollment permission from the patient's hepatologist and monitor values at each study visit. If values increase above 3 times the upper limit of normal, the patient will be discontinued from the study.
  * For patients 1-2 times the upper limit of normal, we will obtain enrollment permission from the patient's physician and monitor per request of the physician.
* Patients with severe or end stage renal disease, defined as a GFR < 15 ml/min or on dialysis
* Patients with a recent (≤ 12 months) history of seizures.
* Patients with uncontrolled narrow-angle glaucoma.
* Patients who have been treated with an experimental agent within the last three months.

Min Age: 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2011-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne C Lee, MD, MMSc, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Lee YC, Chibnik LB, Lu B, Wasan AD, Edwards RR, Fossel AH, Helfgott SM, Solomon DH, Clauw DJ, Karlson EW. The relationship between disease activity, sleep, psychiatric distress and pain sensitivity in rheumatoid arthritis: a cross-sectional study. Arthritis Res Ther. 2009;11(5):R160. doi: 10.1186/ar2842. Epub 2009 Oct 29. PMID 19874580
- [Derived] Lee YC, Massarotti E, Edwards RR, Lu B, Liu C, Lo Y, Wohlfahrt A, Kim ND, Clauw DJ, Solomon DH. Effect of Milnacipran on Pain in Patients with Rheumatoid Arthritis with Widespread Pain: A Randomized Blinded Crossover Trial. J Rheumatol. 2016 Jan;43(1):38-45. doi: 10.3899/jrheum.150550. Epub 2015 Dec 1. PMID 26628607

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 49 patients signed the informed consent document. 8 patients did not meet inclusion criteria and failed screening. 41 patients were randomized and received >= 1 dose of the study drug/placebo. Seven patients stopped participation due to adverse events, and 2 were lost to follow-up. 32 patients completed the study and were analyzed.
Groups:
- Milnacipran and Then Placebo: Participants first received 6 weeks of milnacipran (titrated up to full dose of 50 mg twice daily). This was followed by a 3-week wash-out. Participants then received 6 weeks of placebo.
- Placebo and Then Milnacipran: Participants first received 6 weeks of placebo. This was followed by a 3-week wash-out. After the wash-out period, participants then received 6 weeks of milnacipran (titrated up to full dose of 50 mg twice daily).
Period: First Intervention
Arm/Group | Milnacipran and Then Placebo | Placebo and Then Milnacipran
Started | 23 | 18
Completed | 21 | 17
Not Completed | 2 | 1
Not completed — Adverse Event | 2 | 1
Period: Washout
Arm/Group | Milnacipran and Then Placebo | Placebo and Then Milnacipran
Started | 21 | 17
Completed | 19 | 17
Not Completed | 2 | 0
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Period: 2nd Intervention
Arm/Group | Milnacipran and Then Placebo | Placebo and Then Milnacipran
Started | 19 | 17
Completed | 17 | 15
Not Completed | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: 49 individuals signed the informed consent document. Of these individuals, 8 did not meet inclusion/exclusion criteria. 41 subjects were randomized and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Milnacipran and Then Placebo | Placebo and Then Milnacipran | Total
Number analyzed (Participants) | 23 | 18 | 41
Age, Continuous [Mean (Standard Deviation); unit: Year]
  Age | 56.39 (12.35) | 58.50 (14.79) | 57.32 (13.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 15 | 34
  Male | 4 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Brief Pain Inventory (BPI) Change
Description: A measure of change in scores on the BPI short form, a "24-hr average pain" item, from baseline to 6 weeks, The BPI short form scores ranges from 0-10, with 10 being the worst pain.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Participants who received placebo in either the first or last 6 weeks of the study.
- Milnacipran: Participants who received milnacipran in either the first or last 6 weeks of the study.
  Milnacipran is taken orally. Participants will gradually be increased to a target dose of 50 mg twice daily.
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 5.2 (2.1) | 5.6 (2.0)
  6 weeks | 4.9 (2.1) | 4.8 (2.2)
  Change | -0.3 (2.0) | -0.7 (1.7)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; The difference between the change measured during placebo versus the change during milnacipran treatment. Calculated using Wilcoxon signed rank tests; Test type: Superiority or Other; p = 0.42, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; The difference between the change measured during placebo versus the change during milnacipran treatment. Calculated using linear mixed models; Test type: Superiority or Other; p = 0.37, Mixed Models Analysis — Linear mixed models including treatment, crossover period and treatment sequence. Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05

2. Secondary Outcome: Change in Conditioned Pain Modulation (CPM)
Description: CPM is defined as the difference between pain threshold A (measured after a conditioning stimulus activates pathways that inhibit pain) and pain threshold B (measured before the conditioning stimulus is applied). The conditioning stimulus was immersion of the hand in a cold water bath. Pressure pain threshold was assessed at the trapezius muscle initially. Subjects were then instructed to immerse their hand in a water bath for 30 seconds. At 20 seconds, pressure pain threshold at the trapezius was assessed again. We defined the magnitude of subjects' CPM as the difference in pressure pain threshold between baseline and 20 seconds after cold water immersion. This difference was compared to that measured at 6 weeks. The scale for the difference in CPM ranged from 0-11 kg/cm^2, with 0 indicating no change in CPM between 6 weeks and baseline and 11 indicating the maximum possible change. A greater change in CPM between baseline and 6 weeks is indicative of improvements in CPM.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: kg/cm^2
Groups:
- Milnacipran: Participants who received milnacipran in either the first or last 6 weeks of the study.
  Milnacipran: Participants who take Milnacipran twice a day orally dosage was titrated up to target dosage of 50 mg (12.5 mg, 25 mg and 50 mg).
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
kg/cm^2
  Baseline | 0.8 (1.0) | 0.8 (1.1)
  6 Weeks | 0.9 (1.3) | 0.9 (1.1)
  Change | 0.1 (1.2) | 0.1 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; The difference between the change measured during placebo versus the change during milnacipran treatment. Calculated using the Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.39, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.96, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Symptom Intensity Scale (SIS)
Description: A measure of the change in SIS score from baseline to 6 weeks. The SIS score ranges from 0-9.75, with high scores being worse indicating more widespread pain and fatigue.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Milnacipran: Participants who received milnacipran in either the first or last 6 weeks of the study.
  Milnacipran: Milnacipran comes in 50 mg tablets and is taken orally. Participants will gradually be increased to a target dose of 50 mg twice daily.
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
units on a scale
  Baseline | 5.1 (2.1) | 5.2 (2.0)
  6 weeks | 4.3 (2.4) | 4.5 (8.3)
  Change | -0.8 (1.9) | -0.7 (1.6)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; The difference between the change measured during placebo versus the change during milnacipran treatment. Calculated using Wilcoxon signed-rank tests; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.83, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Thumbnail Pain Threshold
Description: A measure of the change in thumbnail pain threshold from baseline to 6 weeks. Thumbnail pain threshold was determined by applying pressure to a subjectt's thumbnail until the subject felt pain. The difference between the average thumbnail pain threshold (an average for the right and left thumbs) at baseline was compared to that at 6 months. Pain threshold was measured in kg/cm^2. The difference in threshold could range from 0-11 kg/cm^2. A higher difference between thresholds indicates improved pain sensitivity.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
kg/cm^2
  Baseline | 5.8 (3.0) | 5.3 (2.7)
  6 weeks | 5.8 (2.8) | 6.0 (2.8)
  Change | -0.02 (1.4) | 0.7 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.04, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.04, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Trapezius Pain Threshold
Description: A measure of the change in trapezius pain threshold from baseline to 6 weeks. Trapezius pain threshold was determined by applying pressure to a subject's trapezius muscle until the subject felt pain. The difference between the average trapezius pain threshold (an average for the right and left trapezii) at baseline was compared to that at 6 months. Pain threshold was measured in kg/cm^2. The difference in threshold could range from 0-11 kg/cm^2. A higher difference between thresholds indicates improved pain sensitivity.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
kg/cm^2
  Baseline | 4.9 (2.8) | 5.1 (3.1)
  6 Weeks | 5.5 (3.1) | 5.5 (3.1)
  Change | 0.6 (1.5) | 0.4 (1.3)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.89, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.44, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

6. Secondary Outcome: Wrist Pain Threshold
Description: A measure of the change in wrist pain threshold from baseline to 6 weeks. Wrist pain threshold was determined by applying pressure to a subject's wrist until the subject felt pain. The difference between the average wrist pain threshold (an average for the right and left wrists) at baseline was compared to that at 6 months. Pain threshold was measured in kg/cm^2. The difference in threshold could range from 0-11 kg/cm^2. A higher difference between thresholds indicates improved pain sensitivity.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
kg/cm^2
  Baseline | 5.3 (2.7) | 5.0 (2.4)
  6 weeks | 5.9 (3.0) | 5.9 (2.9)
  Change | 0.6 (1.6) | 0.9 (1.5)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.35, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.34, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

7. Secondary Outcome: Knee Pain Threshold
Description: A measure of the change in knee pain threshold from baseline to 6 weeks. Knee pain threshold was determined by applying pressure to a subject's knee until the subject felt pain. The difference between the average knee pain threshold (an average for the right and left knees) at baseline was compared to that at 6 months. Pain threshold was measured in kg/cm^2. The difference in threshold could range from 0-11 kg/cm^2. A higher difference between thresholds indicates improved pain sensitivity.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: kg/cm^2
Arm/Group | Placebo | Milnacipran
Number analyzed (Participants) | 32 | 32
kg/cm^2
  Baseline | 7.0 (3.1) | 6.9 (3.2)
  6 weeks | 7.3 (3.1) | 7.3 (3.2)
  Change | 0.3 (1.8) | 0.3 (1.4)
Statistical Analysis 1: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.72, Wilcoxon (Mann-Whitney) — Not adjusted for multiple comparisons. A priori threshold for statistical significance was < 0.05
Statistical Analysis 2: Comparison: Placebo vs Milnacipran; [analysis description as in outcome 1, analysis 2]; Test type: Superiority or Other; p = 0.82, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: 6 weeks for intervention with a period of 3 weeks of washout between each intervention period.
Groups:
- Milnacipran: Participants received milnacipran for 6 weeks. The dose was titrated according to the following schedule: 1) Days 1-3: milnacipran 12.5 mg twice daily, 2) Days 4-6: milnacipran 25 mg twice daily, 3) Days 7-42: milnacipran 50 mg twice daily. If participants could not tolerate the full dose, the dose was decreased to the highest tolerated dose.
- Placebo: Participants received placebo tablets for 6 weeks. The tablets were identical in appearance to the milnacipran tablets.
- Washout Period: This 3-week period occurred after the first 6 weeks (when participants either received milnacipran or placebo). During the washout period, participants down titrated from the full dosage of milnacipran/placebo to nothing.
Arm/Group | Milnacipran | Placebo | Washout Period
Serious Adverse Events (participants affected / at risk) | 0/41 | 1/41 | 0/41
Other Adverse Events (participants affected / at risk) | 17/41 | 8/41 | 1/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=41) | Placebo (N=41) | Washout Period (N=41)
Colon Abscess (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Milnacipran (N=41) | Placebo (N=41) | Washout Period (N=41)
Headache (General disorders) | 2 (2) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 11 (12) | 3 (4) | 1 (1)
Dizziness (General disorders) | 2 (2) | 1 (2) | 1 (1)
Sleep Problems (General disorders) | 3 (3) | 2 (2) | 0 (0)
Loss of appetite (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Urinary Hesitation (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0)
Parathesthesias (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No